CLINICAL TRIAL: NCT03662971
Title: Phase I Clinical Trial to Evaluate the Tolerance, Safety and Pharmacokinetics of Germinal Peptide Eye Drops in Healthy Volunteers
Brief Title: Evaluate the Tolerance, Safety and Pharmacokinetics of Germinal Peptide Eye Drops in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhaoke (Guangzhou) Ophthalmology Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZK-SFT-201704
Record Dates: First submitted 2018-08-28; First posted 2018-09-10 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2019-05

CONDITIONS: Corneal Defect

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- 0.0005% single-dose (Experimental): Two subjects will be treated with Germinal peptide eye drops 0.0005% single dose.
  Interventions: Drug: Germinal peptide eye drops
- 0.001% single-dose (Experimental): Ten subjects will be treated with Germinal peptide eye drops 0.001% single dose (eight treatment and two placebo).
  Interventions: Drug: Germinal peptide eye drops
- 0.002% single-dose (Experimental): Ten subjects will be treated with Germinal peptide eye drops 0.002% single dose (eight treatment and two placebo).
  Interventions: Drug: Germinal peptide eye drops
- 0.004% single-dose (Experimental): Ten subjects will be treated with Germinal peptide eye drops 0.004% single dose (eight treatment and two placebo).
  Interventions: Drug: Germinal peptide eye drops
- 0.008% single-dose (Experimental): Ten subjects will be treated with Germinal peptide eye drops 0.008% single dose (eight treatment and two placebo).
  Interventions: Drug: Germinal peptide eye drops
- 0.002% multiple-dose (Experimental): Ten subjects will be treated with Germinal peptide eye drops 0.002% multiple dose (eight treatment and two placebo).
  Interventions: Drug: Germinal peptide eye drops
- 0.004% multiple-dose (Experimental): Ten subjects will be treated with Germinal peptide eye drops 0.004% multiple dose (eight treatment and two placebo).
  Interventions: Drug: Germinal peptide eye drops
- 0.008% multiple-dose (Experimental): Ten subjects will be treated with Germinal peptide eye drops 0.008% multiple dose (eight treatment and two placebo).
  Interventions: Drug: Germinal peptide eye drops

INTERVENTIONS:
Drug: Germinal peptide eye drops — Germinal peptide eye drops of 0.0005%, 0.001%, 0.002%, 0.004% and 0.008%
  Other Names: Germinal peptide

SUMMARY:
Phase I Clinical Trial to Evaluate the Tolerance, Safety and Pharmacokinetics of Germinal Peptide Eye Drops in Healthy Volunteers.

DETAILED DESCRIPTION:
The subjects enrolled in this study are healthy volunteers, divided into single dose groups and multiple doses groups with dose escalation.The study is designed to assign the subjects to five single-dose groups from low to high (0.0005%, 0.001%, 0.002%, 0.004% and 0.008%), and three multiple-dose groups (0.002%, 0.004% and 0.008%), with both male and female subjects in each group. This clinical trial is a double-blind design.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers aged between 18 and 45, both male and female;
2. The body mass index was between 19 and 26kg/m2 (including the critical value), the weight of male ≥50kg, and that of female ≥45kg；
3. The BCVA of both eyes should be ≥ 1.0, and the intraocular pressure, slit lamp and fundus examination were all normal or abnormal values without clinical significance；
4. Before the test, physical examination, vital signs, ECG, laboratory examination were in the normal range or no clinical significance；
5. Women of childbearing age have negative blood pregnancy test, the subject should ensure that effective contraceptive measures are taken within 1 month before inclusion, and the subject (including male ) is willing to have no pregnancy plan in the next 6 months and voluntarily take effective contraceptive measures;
6. Subjects volunteered to participate in the study and signed ICF.

Exclusion Criteria:

1. Patients with eye diseases, including a history of internal eye surgery or laser surgery;
2. History of central nervous system, spirit system, cardiovascular system, kidney system, liver system, respiration system, metabolism and skeletal muscle system;
3. Positive results of hepatitis B virus surface antigen (HBsAg), anti-hepatitis C virus (HCV) antibodies , syphilis spiral antibody (TP-Ab) or r anti-human immunodeficiency virus (HIV) antibodies;
4. A significant clinical history of allergic reactions, especially drug allergies, especially allergic to any ingredient in Germinal peptide eye drops;
5. Smoking more than 5 cigarettes a day on average;
6. Suspicion or actual alcohol dependence; intake of more than 2 units of alcohol per day on average in 3 months (1 unit =10 mL ethanol,, 1 unit =200mL of beer or 25 mL of spirits with 40% alcohol or 83 mL of wine with 12% alcohol) or alcohol test positive;
7. History of drug abuse, or a positive urine test of ketamine, morphine, methamphetamine, dimethylamine and tetrahydrocannabinoid;
8. Take any medicine within 2 weeks before screening;
9. Participated in clinical trials within 3 months before screening;
10. Donation or loss of more than 400 ml of blood within 3 months before screening
11. Used ophthalmic drugs or eyelash growth fluid within 2 weeks before screening;
12. Used contact lenses or cosmetic contact lenses within 2 weeks before screening;
13. Pregnant or lactating women and planned pregnancies (including male subjects);
14. The researcher considers that it is not suitable for the trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2018-12-04 (Actual); Study Completion 2019-10-24 (Actual)

PRIMARY OUTCOMES:
ocular symptoms | Within two days after administration
  Ocular signs: conjunctival congestion, corneal epithelial injury, conjunctival edema, anterior chamber glow.

SECONDARY OUTCOMES:
Area under curve （0-t） | Within two days after administration
  AUC（0-t）
Area under curve（0-∞） | Within two days after administration
  AUC（0-∞）
Peak concentration | Within two days after administration
  Cmax
Peak time | Within two days after administration
  Tmax
Half life | Within two days after administration
  t1/2
Apparent volume of distribution | Within two days after administration
  Vd
Elimination rate constant | Within two days after administration
  Kel
Mean residence time | Within two days after administration
  MRT
Clearance | Within two days after administration
  CL or CL/F
slit lamp examination | Within two days after administration
  Examination of cornea, conjunctiva, sclera, lens and vitreous body.
fundus examination | Within two days after administration
  Observe the change of fundus.
intraocular pressure | Within two days after administration
  Observe the change of intraocular pressure.
vision | Within two days after administration
  Observe the change of vision.
12-lead ECG | Within two days after administration
  Observe the change of 12-lead ECG.
AE | Within two days after administration
  Observe the occurrence and record of AE.
corneal fluorescein staining | Within two days after administration
  Observe the change of corneal fluorescein staining.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zhao, PhD, Study Director — Beijing Tongren Hospital
Locations (1):
- Xiuli Zhao, Beijing, China

IPD SHARING:
Plan to Share IPD: No